CLINICAL TRIAL: NCT03275441
Title: Investigation of a Protocol Change (Shorter Dark-adaptation) on the Electroretinogram (ERG) in an Adult Patient Population (SHERG)
Brief Title: Electroretinography: Investigation of a Protocol Change
Acronym: SHERG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN17OP146
Record Dates: First submitted 2017-03-22; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Dark-adapted ERG
Keywords: electroretinogram; ERG; dark-adaptation; ophthalmology; electrophysiology; ISCEV; electroretinography; scotopic
MeSH Terms: interventions — Electroretinography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients: Adult patients attending hospital for clinical visual electrophysiology.
  Interventions: Diagnostic Test: Electroretinography

INTERVENTIONS:
Diagnostic Test: Electroretinography — An additional electroretinogram performed after 10 minutes of dark adaptation.

SUMMARY:
The study evaluates whether an eye test called an electroretinogram (ERG) can be shortened and still produce the same diagnostic results. The results of this study may allow test times to be reduced which will have benefits such as improved patient compliance during shorter testing and increased clinic efficiency.

DETAILED DESCRIPTION:
A full-field electroretinogram (ERG) is a standardised eye test undertaken in specialist hospital clinics. ERGs are useful for diagnosing and monitoring retinal diseases. The retina is stimulated by showing patients flashes of light and the resulting electrical response from the eye is recorded using delicate electrodes that touch the surface of the eye. For the first section of the test, patient's eyes are allowed to adjust to the dark to ensure the parts of the retina responsible for seeing in dimly-lit conditions are being tested.

The international ERG Standard says patients must sit in the dark for 20 minutes. The investigators have evidence to suggest the test may be equally useful after only 10 minutes in the dark. The investigators plan to compare ERGs recorded from patients who have spent only 10 minutes in the dark with ERGs recorded from the same patients after the full 20 minutes in the dark. If the difference is suitably small, as found in a preliminary study of healthy individuals, it could be justifiable to shorten the routine patient protocol.

Subjects for this study will be recruited from the adult population routinely attending for an outpatient ERG test. During their routine ERG test, 10 minutes into the 20 minute wait in the dark, the investigators propose recording an additional, identical set of ERG tests. This will not add extra time to the clinical test.

Participants will not need any follow-up for the research study. The study requires 262 patients to test the hypothesis, and the investigators estimate this will take about 5-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the adult visual electrophysiology service regardless of clinical condition, and who require dark-adapted electroretinography as part of their appointment
* Male or female
* All ethnicities

Exclusion Criteria:

* Patients less than 18 years old
* Patients who might have difficulties understanding the participant information provided (for example, those patients requiring a translator, or who have learning difficulties)
* Patients with photosensitive epilepsy
* Patients appointed for clinical testing urgently, or via telephone, who will not have had an opportunity to receive and review the participant information sheet ahead of the clinical appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient population attending hospital for routine clinical electroretinography.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Rate of classification for ERG following 10 minute dark adaptation | (During first & only study visit) Dark-adapted ERG test following 10 minutes of dark adaptation
  The rate of classification (normal vs abnormal) for testing conducted after 10 minutes of dark adaptation.
Rate of classification (normal vs abnormal) for ERG following 20 minute dark adaptation | (During first & only study visit) Dark-adapted ERG test following 20 minutes of dark adaptation
  The rate of classification (normal vs abnormal) for testing conducted after 20 minutes of dark adaptation.

SECONDARY OUTCOMES:
Response amplitude after 10 minutes | (During first & only study visit) Dark-adapted ERG test following 10 minutes of dark adaptation
  Measurement of the amplitude of responses following 10 minutes of dark adaptation.
Response amplitude after 20 minutes | (During first & only study visit) Dark-adapted ERG test following 20 minutes of dark adaptation
  Measurement of the amplitude of responses following 20 minutes of dark adaptation.
Response timing | (During first & only study visit) Dark-adapted ERG test following 10 minutes of dark adaptation
  Measurement of the amplitude of responses following 10 minutes of dark adaptation.
Response timing | (During first & only study visit) Dark-adapted ERG test following 20 minutes of dark adaptation
  Measurement of the amplitude of responses following 20 minutes of dark adaptation.
Response variability | (During first & only study visit) Dark-adapted ERG test following 10 minutes of dark adaptation
  Measurement of the variability of responses following 10 minutes of dark
Response variability | (During first & only study visit) Dark-adapted ERG test following 20 minutes of dark adaptation
  Measurement of the variability of responses following 20 minutes of dark

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Hamilton, PhD, Study Director — NHS Greater Glasgow & Clyde; Kirsten Graham, MSc, Principal Investigator — NHS Greater Glasgow & Clyde; Richard Hagan, PhD, Principal Investigator — NHS Royal Liverpool University Hospital

IPD SHARING:
Plan to Share IPD: No